CLINICAL TRIAL: NCT05757258
Title: Cardiovascular Biomarkers in Diabetic Patients Undergoing Endovascular Revascularization for Chronic Limb-threatening Ischemia (CLTI).
Brief Title: Cardiovascular Biomarkers in Peripheral Artery Disease.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Flex Andrea, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2012
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Artery Disease
Keywords: Cytokines; MACE; MALE; Atherosclerosis; Diabetes mellitus; Peripheral artery disease
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the best medical management, many patients with peripheral artery disease (PAD) who undergo lower extremity endovascular revascularization experience adverse cardiovascular outcomes and postoperative complications that may increase the risk of acute limb ischemia or amputation. There are no clear molecular associations that could explain the differences in outcomes after endovascular therapy in patients with PAD. The variable outcomes following endovascular therapy may depend, at least in part, on the profile of cytokines involved in inflammatory and atherosclerotic processes.

The goal of this observational study is to evaluate the potential use of circulating IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 levels as biomarkers of major adverse limb events (MALE) and major adverse cardiovascular events (MACE) in diabetic patients with PAD and chronic limb-threatening ischemia (CLTI) requiring a procedure of endovascular revascularization.

The main questions it aims to answer are:

* association between serum levels of IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 at baseline and major adverse limb events (MALE) after lower extremity revascularization.
* association between serum levels of IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 at baseline and major adverse cardiovascular events (MACE) after lower extremity revascularization.

Diabetic patients with CLTI requiring lower extremity endovascular revascularization will undergo blood sampling for the dosage of circulating IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 before the endovascular procedure.

Incidence of MALE and MACE will be collected in a 12-months follow-up and will be associated with IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years
* diagnosis of T2DM present for a least one year
* Ankle/Brachial Index (ABI) of less than 0.80
* lower limb stenosis greater than 50% documented by Ultrasound Color Doppler (US)
* category 4 or 5 of PAD in accordance with the Rutherford classification
* presence of CLTI requiring endovascular treatment

Exclusion Criteria:

* pregnancy
* acute infections at present or in the previous month
* diabetic foot ulcers with sign of infection or osteomyelitis
* previous lower-limb endovascular or surgical revascularization within the past 3 months
* diabetic peripheral neuropathy
* liver disease with a functional status B or C in accord to Child-Pugh classification
* congenital or acquired thrombophilia
* active autoimmune disease
* active cancer
* organ transplantation
* life expectancy < 12 months
* contraindication to antiplatelet therapy
* contraindication to endovascular revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll consecutive patients with type 2 diabetes mellitus and PAD needing lower extremity and admitted to Internal Medicine Cardiovascular Unit of the Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma.
Sampling Method: Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Association between incidence of MALE and IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels | 12-months follow-up
  To evaluate the association between IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels before endovascular revascularization and incidence of MALE during the follow-up period.

SECONDARY OUTCOMES:
Association between incidence of myocardial infarction and IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels | 12-months follow-up
  To evaluate the association between IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels before endovascular revascularization and incidence of myocardial infarction during the follow-up period.
Association between incidence of stroke and IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels | 12-months follow-up
  To evaluate the association between IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels before endovascular revascularization and incidence of stroke during the follow-up period.
Association between incidence of cardiovascular death and IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels | 12-months follow-up
  To evaluate the association between IL-1, IL-6, TNF-alpha, C reactive protein, HMGB-1, osteoprotegerin, sortilin and omentin-1 serum levels before endovascular revascularization and incidence of cardiovascular death during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Flex, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy